CLINICAL TRIAL: NCT01640808
Title: NIK-333(Peretinoin) PhaseⅢ Study Investigation of the Efficacy and Safety to Suppress Recurrence of Hepatitis C Virus(HCV)-Positive Hepatocellular Carcinoma(HCC), Multicenter, Randomised, Double-blind, Placebo-controlled, Parallel-group Study
Brief Title: Study of Peretinoin for Suppressing Recurrence of HCV-positive HCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NIK-333-05
Record Dates: First submitted 2012-07-10; First posted 2012-07-16 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Hepatic Neoplasm Malignant Recurrent

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- NIK-333(peretinoin) (Experimental)
  Interventions: Drug: NIK-333(peretinoin)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NIK-333(peretinoin) — 600mg (8 x 75mg capsules) orally, twice a day
  Arms: NIK-333(peretinoin)
Drug: Placebo — Placebo (8 x Placebo capsules) orally, twice a day
  Arms: Placebo

SUMMARY:
The purpose of this study is to verify the superiority of NIK-333 (Peretinoin) to placebo in inhibiting the recurrence of HCV-positive HCC in patients showing complete cure of the disease, with the recurrence-free survival as the primary endpoint, in a multi-center, randomized, double-blind, placebo-controlled, parallel-group comparison study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HCV-positive HCC who meet the following conditions before radical treatment

   * Patients diagnosed as having typical HCC on dynamic CT,CTA/CTAP, or dynamic MRI (nodule visualized as a high signal intensity area in the arterial phase and as a relatively low signal intensity area in the portal and equilibrium phases) performed within 8 weeks (56 days) before treatment start prior to radical therapy
   * Patients with the first primary HCC or the first recurrence of primary HCC
2. Patients who received the radical therapies. The treatment duration (from the start to the end of the treatment) should be within 4 weeks (28 days) for each of the radical therapies.
3. Patients showing a complete cure, as confirmed by the dynamic CT images taken from 8 weeks (56 days) to 12 weeks (84 days) after the end of the treatment show a non-stained low-concentration area overlapping the tumor image observed before complete cure.
4. Patients who are able to begin treatment with the study drug within 8 weeks (56 days) after dynamic CT to confirm complete cure
5. Patients confirmed of satisfying the following conditions based on the screening performed at subject registration

   * Positive for serum hepatitis C virus nucleic acid (HCV-RNA)
   * Grade A on Child-Pugh classification
   * Platelet count of 50 000/µL or higher
6. Patients with ECOG Performance Status score of 0 to 1
7. Patients of the age of 20 years or older at the time of informed consent

Exclusion Criteria:

1. Patients positive for HBs antigen
2. Patients showing vascular invasion of HCC on imaging diagnosis
3. Patients who have also undergone transcatheter arterial embolization therapy (TAE/TACE), transarterial infusion therapy (TAI), and chemolipiodolization in combination with the radical therapy
4. 4 Patients who want to receive antiviral therapy such as concomitant therapy with intaferon during the study period
5. Patients who have received other study drugs, anticancer drugs, or interferons after radical therapy
6. Patients who have hypertension as a complication, and whose blood pressure cannot be controlled by drug therapy (systolic blood pressure of 160 mmHg or higher or diastolic blood pressure of 100 mmHg or higher, as determined at subject registration)
7. Patients who have a history of allergy to CT contrast media, and whose participation in this study is judged to be inappropriate by the investigator or the subinvestigator
8. Patients with a history of total gastrectomy
9. Patients with a history of cardiac arrest
10. Patients with any of the following laboratory values or complications

    * Creatinine>= 1.5mg/dL
    * Albumin urine >= 1000mg/g Creatinine
    * Cardiac disorder corresponding to CTC-AE grade 3 in severity
    * HbA1c >= 7.4 under treatment with insulin
    * Autoimmune disease or asthma being treated with oral steroid
11. Patients confirmed of having another malignant neoplasm or who had undergone a radical therapy of HCC within the past 5 years to treat another malignant neoplasm (however, this does not apply to endoscopic resection and resection of intraepithelial carcinoma)
12. Patients who are pregnant, who have a possibility of being pregnant or who have a desire to become pregnant during the study period
13. Lactating women
14. Patients who have a history of allergy to retinoid-related substances (vitamin A, etc.) in the past
15. Patients who participated in another clinical study within past 6 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- Japan (51):
  - Nagoya, Aichi-ken
  - Kashiwa, Chiba
  - Matsuyama, Ehime
  - Iizuka, Fukuoka
  - Kurume, Fukuoka
  - Ōgaki, Gifu
  - Sapporo, Hokkaido
  - Himeji, Hyōgo
  - Kobe, Hyōgo
  - Nishinomiya, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Kawasaki, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Nankoku, Kochi
  - Kurashiki, Okayama-ken
  - Ikeda, Osaka
  - Moriguchi, Osaka
  - Sakai, Osaka
  - Sayama, Osaka
  - Suita, Osaka
  - Iruma, Saitama
  - Sunto-gun, Shizuoka
  - Shimotsuke, Tochigi
  - Bunkyo-ku,, Tokyo
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Chuo-ku, Tokyo
  - Minato-ku, Tokyo
  - Musashino, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shibuya-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Shimonoseki, Yamaguchi
  - Ube, Yamaguchi
  - Kofu, Yamanashi
  - Chiba
  - Fukuoka
  - Gifu
  - Hiroshima
  - Kagoshima
  - Kumamoto
  - Nagasaki
  - Niigata
  - Okayama
  - Osaka
  - Ōita
  - Saga
  - Tokushima
  - Wakayama

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screened:778 Enrolled:616 Received treatment:610
Period: Overall Study
Arm/Group | NIK-333(Peretinoin) | Placebo
Started | 309 | 307
Subjects Received Treatment | 305 | 305
Completed | 251 | 291
Not Completed | 58 | 16
Not completed — Unable to continue dynamic CT | 14 | 4
Not completed — Withdrawal by Subject | 12 | 4
Not completed — Lost to Follow-up | 4 | 0
Not completed — Start an antiviral therapy using IFN | 3 | 0
Not completed — Administration of anticancer drugs | 2 | 1
Not completed — Physician Decision | 19 | 5
Not completed — Randomized but not treated | 4 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) consisted of 605 subjects among 616 randomized subjects. Reasons for 11 excluded subjects are as following;
  * 6 Subjects (NIK-333 group: 4, Placebo group: 2) who did not take any study drugs
  * 5 Subjects (NIK-333 group: 4, Placebo group: 1) who had no efficacy data
Groups:
- Total: Total of all reporting groups
Arm/Group | NIK-333(Peretinoin) | Placebo | Total
Number analyzed (Participants) | 301 | 304 | 605
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 51 | 44 | 95
  Between 65 and 75 years | 100 | 124 | 224
  >=75 years | 150 | 136 | 286
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 123 | 241
  Male | 183 | 181 | 364

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival
Description: HCC recurrence was defined as the appearance of new intrahepatic lesions which was confirmed based on findings of hypervascularity (nodules enhanced in the arterial phase and washout in the late phase) by dynamic CT images, or a new extrahepatic metastasis. Recurrence of intrahepatic HCC was evaluated by an independent image reading committee.
  RFS was defined as the time from randomization to HCC recurrence or death from any cause, whichever occurred first. For subjects who terminated the study without HCC recurrence or death, RFS was censored at the day of the latest dynamic CT examination.
Time Frame: Date of randomization to the date of recurrence of HCC (followed every 12 weeks) or death (whichever occurs first)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | NIK-333(Peretinoin) | Placebo
Number analyzed (Participants) | 301 | 304
Days | 809.0 [650.0 to 1026.0] | 751.0 [600.0 to 928.0]
Statistical Analysis 1: Comparison: NIK-333(Peretinoin) vs Placebo; Test type: Superiority; p = 0.351, Log Rank — A two-sided significance level was set at 0.05. Adjustment of multiplicity considering interim analysis is conducted by the Lan DeMets' method of α consumption function; Hazard Ratio (HR) = 0.900, 95% CI 2-sided [0.720 to 1.124]

2. Secondary Outcome: Disease-free Survival
Description: DFS was defined as the time from randomization to HCC recurrence, death from any cause or occurrence of secondary cancer (malignant tumors other than HCC), whichever occurred first. For subjects who terminated the study without HCC recurrence, death, or occurrence of secondary cancer, DFS was censored at the day of the latest dynamic CT examination.
Time Frame: Date of randomization to the date of recurrence of HCC (followed every 12 weeks), death, or secondary cancer (malignant tumors other than HCC)(whichever occurs first)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | NIK-333(Peretinoin) | Placebo
Number analyzed (Participants) | 301 | 304
Days | 686.0 [532.0 to 860.0] | 642.0 [528.0 to 771.0]
Statistical Analysis 1: Comparison: NIK-333(Peretinoin) vs Placebo; Test type: Superiority; p = 0.222, Log Rank — A two-sided significance level was set at 0.05; Hazard Ratio (HR) = 0.875, 95% CI 2-sided [0.706 to 1.085]

3. Secondary Outcome: Time to Recurrence
Description: TTR was defined as the time from randomization to HCC recurrence. For subjects who terminated the study without HCC recurrence, TTR was censored at the day of the latest dynamic CT examination.
Time Frame: Date of randomization to the date of recurrence of HCC(followed every 12 weeks)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | NIK-333(Peretinoin) | Placebo
Number analyzed (Participants) | 301 | 304
Days | 842.0 [673.0 to 1094.0] | 764.0 [608.0 to 936.0]
Statistical Analysis 1: Comparison: NIK-333(Peretinoin) vs Placebo; Test type: Superiority; p = 0.279, Log Rank — A two-sided significance level was set at 0.05; Hazard Ratio (HR) = 0.882, 95% CI 2-sided [0.703 to 1.108]

ADVERSE EVENTS:
Time Frame: From the starting day of study drug administration to 35 days after the discontinuation of the study drug administration, up to approximately 4.3 years.
Description: Safety analysis set consisted of 610 subjects who received treatment. Since the number of SAE of HCC recurrence is larger than other SAEs and is greater in the Placebo group than in NIK-333 group, we consider that there is a concern of underestimating the safety issue from the following points.
  * It becomes difficult to understand what extent SAE that pose a safety concern have occurred.
  * The incidence of SAE in placebo group and NIK-333 group appears to be similar.
Arm/Group | NIK-333(Peretinoin) | Placebo
Serious Adverse Events (participants affected / at risk) | 222/305 | 223/305
Other Adverse Events (participants affected / at risk) | 253/305 | 193/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NIK-333(Peretinoin) (N=305) | Placebo (N=305)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 2 (3) | 0 (0)
Blepharochalasis (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 7 (7)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 16 (16) | 4 (4)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 3 (3)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric varices (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 4 (4) | 4 (4)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 8 (8) | 7 (10)
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal varices (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 2 (2)
Drowning (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Performance status decreased (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Implant site haematoma (General disorders) | 1 (1) | 0 (0)
Disuse syndrome (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 2 (3)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (3)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 2 (2) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (6) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 6 (7) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heat illness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Gastric cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Gastric cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (3)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 3 (3) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 2 (3)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 3 (3) | 3 (3)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 7 (8) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 131 (131) | 171 (171)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NIK-333(Peretinoin) (N=305) | Placebo (N=305)
Ascites (Gastrointestinal disorders) | 41 (42) | 12 (14)
Constipation (Gastrointestinal disorders) | 35 (39) | 24 (24)
Diarrhoea (Gastrointestinal disorders) | 34 (41) | 28 (32)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 22 (22) | 6 (6)
Oedema peripheral (General disorders) | 40 (42) | 22 (26)
Pyrexia (General disorders) | 21 (25) | 16 (17)
Hepatic function abnormal (Hepatobiliary disorders) | 16 (16) | 14 (16)
Cystitis (Infections and infestations) | 32 (45) | 14 (20)
Nasopharyngitis (Infections and infestations) | 109 (167) | 99 (187)
Contusion (Injury, poisoning and procedural complications) | 25 (27) | 13 (13)
Albumin urine present (Investigations) | 21 (22) | 5 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (19) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (20) | 14 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 38 (40) | 17 (17)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 (13) | 16 (18)
Headache (Nervous system disorders) | 18 (19) | 18 (23)
Insomnia (Psychiatric disorders) | 24 (24) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 17 (27)
Nail disorder (Skin and subcutaneous tissue disorders) | 20 (20) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 27 (29) | 33 (38)
Rash (Skin and subcutaneous tissue disorders) | 17 (18) | 13 (16)
Hypertension (Vascular disorders) | 95 (100) | 30 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No